CLINICAL TRIAL: NCT03701581
Title: 4-aminopyridine Treatment for Nerve Injury Resulting From Radical Retro-Pubic Prostatectomy
Brief Title: 4-aminopyridine Treatment for Nerve Injury
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: John Elfar (Other)
Responsible Party: Sponsor-Investigator, John Elfar, Tenured Professor, Chairman, Department of Orthopaedic Surgery, University of Arizona
Organization: University of Arizona (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 00003869
Record Dates: First submitted 2017-10-25; First posted 2018-10-10 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Nerve Injury; Prostate Cancer
Keywords: prostatectomy; erectile dysfunction; prostate cancer; nerve injury; incontinence
MeSH Terms: conditions — Prostatic Neoplasms; Erectile Dysfunction | interventions — 4-Aminopyridine

STUDY DESIGN:
Intervention Model Description: Randomized placebo-controlled trial of 4AP vs placebo for nerve injury
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group A: Investigational Treatment (Experimental): * FDA-approved 10mg dalfampridine (generic Ampyra)
  * Subjects will not take more than 2 tablets in a 24-hour period
  * Subjects will take the tablets whole. They will not break, crush, chew, or dissolve tablets before swallowing.
  * The subjects will be told that the medication is released slowly over time and if the tablet is broken, the medicine may be released too fast which can raise the chance of having a seizure.
  * Study drug can be taken with or without food.
  * If a dose is missed they should not make up the missed dose. They will be told not to take two doses at the same time but to take the next dose at the regular scheduled time.
  * Subjects will be reminded not to take study drug together with other aminopyridine medications, including compounded 4-AP (sometimes called 4-aminopyridine or fampridine).
  Interventions: Drug: 4-Aminopyridine
- Group B: Placebo (Placebo Comparator): Subjects will receive an oral dose of placebo treatment the day after surgery, continuing daily for 2 months (60 days) following the same administration instructions as the investigational treatment. The placebo tablets will be manufactured by a licensed compounding pharmacy. The Investigational Drug Service at Banner University Medical Center will manage the placebos.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: 4-Aminopyridine — FDA-approved tablets.
  Other Names: 4-AP; Fampridine; Dalfampridine
  Arms: Group A: Investigational Treatment
Other: Placebo — Placebo will be tooled to look similar to the study drug.
  Arms: Group B: Placebo

SUMMARY:
To evaluate the role of 4-aminopyridine (4-AP) on the course of recovery after peripheral nerve traction and/or crush injury. This study aims to test the hypothesis that 4-aminopyridine speeds the often slow and unpredictable recovery after peripheral nerve traction and/or crush injuries.

DETAILED DESCRIPTION:
To evaluate the role of 4-AP on the recovery of nerve function we will be giving patients with prostate cancer who are undergoing robot assisted radical prostatectomy (RP) either 4-AP or placebo in the perioperative period. This population of patients was selected as nerve crush injury during RP is thought to contribute to erectile dysfunction and urinary continence post operatively.

ELIGIBILITY:
Inclusion Criteria

* Male patients with organ-confined, non-metastatic prostate cancer (stages cT1c-T2c), planning to undergo Robotic-Assisted Laparoscopic Bilateral Nerve Sparing Radical Prostatectomy (NSRP)
* Prostate-Specific Antigen (PSA) levels less than 15 ng/ml (within the last 12 months), with biopsy-proven prostate cancer, for whom postoperative adjuvant therapy (e.g. radiation or androgen deprivation therapy) is not expected to be needed
* Ages 45-75
* An Abridged International Index of Erectile Function-Erectile Function (IIEF-5) score of greater than or equal to 17 at time of screening
* Has experienced at least 6 months of regular sexual activity and sexual activity during the 12 weeks prior to prostate biopsy or surgery
* Willingness to abstain from treatments for Erectile Dysfunction until 3 months after surgery
* Willingness to participate and able to provide informed consent

Exclusion Criteria

* Planned adjuvant therapy after NSRP based on specimen pathology and stage of prostate cancer (stage T3 or greater), positive lymph nodes or positive surgical margins
* Neo-adjuvant therapy prior to NSRP
* History of recurrent prostate cancer
* History of seizures, multiple sclerosis, stroke or any other diagnosed neurological disorder
* History of non-organ confined or metastatic prostate cancer (clinical Stages T3 or greater)
* History of known hypersensitivity to 4AP
* Patients with history of penile surgery other than circumcision or endoscopic urethral stricture surgery
* Renal impairment based on calculated GFR (GFR<60 mL/min)
* Use of any other aminopyridine medications for any other indication

Ages: 45 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Restricted to male subjects due to the inclusion criteria of prostate cancer.
Enrollment: 70 (Estimated)
Dates: Start 2021-06-05 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Michigan Incontinence Sympton Index (M-ISI) (change over time) | Pre-operative visit, and every seven days (starting after surgery, i.e., 7 days post-op) for 6 months (up to 25 times).
  Incontinence measurement (change over time)
International Index of Erectile Function (IIEF) (change over time) | Pre-operative visit, and every seven days (starting after surgery, i.e., 7 days post-op) for 6 months (up to 25 times).
  Erectile function measurement tool. (change over time)
Placebo vs. Active Drug Questionnaire | through study completion, an average of 1 year
  Specific questions regarding patient blinding

SECONDARY OUTCOMES:
Drug Diary | Daily for 90 days.
  Subjects will record the time each day that they take the study drug/ placebo.
Attempted Sexual Activity Questionnaire | Pre-operative visit, and every seven days (starting after surgery, i.e., 7 days post-op) for 6 months (up to 25 times).
  Sexual activity assessment

CONTACTS AND LOCATIONS:
Overall Officials: Rashid Sayyid, MD, Principal Investigator — University of Arizona; John Elfar, MD, Study Chair — University of Arizona
Locations (2):
- United States (2):
  - University of Arizona, Tucson, Arizona
  - University of Rochester, Rochester, New York

IPD SHARING:
Plan to Share IPD: Yes
At the conclusion of the study, de-identified patient outcomes will be provided with publication of results. This includes outcomes data as listed in the primary and secondary outcomes sections.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: For five years post study conclusion and publication.
Access Criteria: Per the accepting journal.

REFERENCES:
- [Derived] Ghazi A, Osinski TL, Feng C, Horne A, Elfar J. 4-Aminopyridine treatment for nerve injury resulting from radical retro-pubic prostatectomy: a single-center double-blind, randomized, placebo-controlled study. Trials. 2024 May 21;25(1):332. doi: 10.1186/s13063-024-08102-z. PMID 38773595